CLINICAL TRIAL: NCT02149680
Title: Long-term Follow-up of Patients Having Had an Epidural Blood Patch Following Accidental Dural Puncture During Labour or Caesarean Section
Brief Title: Long-term Effects of Accidental Dural Puncture in Patients Having Had an Epidural Blood Patch (LEAP)
Acronym: LEAP
Status: Completed | Type: Observational
Sponsor: Örebro University, Sweden (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Anil Gupta, Associate Professor, Örebro University, Sweden
Other Study IDs: LEAP-2013
Record Dates: First submitted 2014-05-25; First posted 2014-05-29 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Post-dural Puncture Headache; Post-dural Puncture Backache
Keywords: Post-dural puncture headache; epidural blood patch; labour analgesia; epidural analgesia
MeSH Terms: conditions — Post-Dural Puncture Headache

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Experimental group: Patient who has had an epidural blood patch following accidental dura puncture during pregnancy
- Control Group: Women in the same group, equal numbers of those with or without epidurals, without accidental dural puncture, similar parity would constitute the control group. They would be chose at random, 10 times the number in the experimental group (n = 600).

SUMMARY:
Accidental dural puncture (ADP) during placement of an epidural catheter for anesthesia and analgesia is a well known complication. Previous studies have found audiometric deterioration following ADP. Epidural blood patch (EBP) is a common method for treating postural headache in patients with accidental dural puncture. In most cases, one-two patches are needed for successful management. Long-term effects of EBP on the incidence of backache, headache and early audiometric deterioration are few or non-existant. The present study aims to determine the long-term sequelae of EDP in parturients who had ADP and were treated with an EBP during the years 2005 - 2011.

DETAILED DESCRIPTION:
A major risk with epidural analgesia (EDA) is accidental dural puncture (ADP). ADP occurs in approximately 1% of all pregnant women receiving EDA in connection with childbirth. Postdural puncture headache (PDPH) is the most common complication after ADP and affects approximately 86% of all mothers with ADP. Headache after ADP may be severe and sometimes affects the interaction between the newborn baby and the mother. The headaches are orthostatic which makes the patient bedridden, and are associated with symptoms such as nausea, vomiting, tinnitus and hearing changes. The symptoms are thought to represent leakage of cerebrospinal fluid (CSF), which in turn leads to reduced CSF volume and intracranial hypotension. These volume changes lead to traction of pain-sensitive intracranial structures. There are no studies in the literature that have either confirmed or visualized CSF leakage after ADP. The diagnosis of PDPH is solely based on clinical examination. There are over 50 different treatment options for PDPH. These treatments can be divided into conservative or invasive. Among others, the conservative treatment options include bed rest, caffeine and various pain medications. Several studies have shown the absence of a definite and curative effect of these treatment options. The most widely used invasive method for management of PDPH is epidural blood patch (EBP). EBP was first introduced in the 60's by applying three ml of the patients' own blood epidurally. Over the years, this volume has increased to at least 15-20 ml on the basis of case reports and studies with small number of participants and without any definite scientific evidence. However, EBP should not be applied sooner than 24 hours after the onset of accidental dura puncture, as the risk of failure is higher. Further studies are required in the literature to confirm the efficacy of EBP.

Additionally, the long term effects of EBP remain either unknown or vaguely understood. Are we treating an acute symptom with an invasive method, not knowing the long term sequelae? Since audiometric changes are known to result following ADP, can these changes persist over a long period of time? Therefore, we are interested in assessing the long term effects of EBP on backache, headache and audiometric changes in parturients who delivered during the years 2005 - 2011.

ELIGIBILITY:
Inclusion Criteria:

* Women in the age group 20-45 years
* Delivered during the years 2005-2011
* Region of Örebro and Stockholm, Sweden

Exclusion Criteria:

* Language difficulty
* Mental inadequacy
* Chronic backache or headache
* Pre-eclampsia during pregnancy
* Previous accidental dural puncture

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women who had delivered during the years 2005 - 2011. Experimental group: 60 patients who had an accidental dura puncture during labour or caesarean section and developed post-dura puncture headache and required an epidural blood patch would constitute the experimental group Contro group: 600 patients, identical to the above except that they had no dura puncture and therefore no post-dural puncture headache
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Audiometric changes | 3 - 8 years after event
  Changes in oto-acoustic emission and tone-audiometry

SECONDARY OUTCOMES:
Headache | During the last month
  Has the patient been affected by persistent or positional headaches, their character and localization
Backache | Last 1 year
  Has the patient had problems with persistent backache that either prevents her from working full time, if there is any radiation of pain, its character and localization

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - University Hospital, Örebro
  - Karolinska Hospital, Stockholm

REFERENCES:
- [Background] Darvish B, Gupta A, Alahuhta S, Dahl V, Helbo-Hansen S, Thorsteinsson A, Irestedt L, Dahlgren G. Management of accidental dural puncture and post-dural puncture headache after labour: a Nordic survey. Acta Anaesthesiol Scand. 2011 Jan;55(1):46-53. doi: 10.1111/j.1399-6576.2010.02335.x. Epub 2010 Oct 29. PMID 21039355